CLINICAL TRIAL: NCT00733577
Title: A Single-blinded Randomized, Placebo-controlled, Staggered-parallel, Escalating-dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral SB756050 Administered for 6 Days to Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Test How SB756050 Affects Subjects With Type 2 Diabetes Mellitus After 6 Days of Dosing.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111829
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; pharmacodynamics; safety; pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 15 mg SB756050 or placebo
  Interventions: Drug: SB756050
- Cohort 2 (Experimental): Planned dose for Cohorts 2 50mg SB756050 or placebo
  Interventions: Drug: SB756050
- Cohort 3 (Experimental): Planned dose for Cohort 3 150mg SB756050 or placebo
  Interventions: Drug: SB756050
- Cohort 4 (Experimental): Planned dose for Cohort 4 600mg SB756050 or placebo
  Interventions: Drug: SB756050

INTERVENTIONS:
Drug: SB756050 — doses are planned to be 15mg to 600mg doses may be altered based on plasma concentrations

SUMMARY:
This is an escalating dose study in subjects with T2DM, which will consist of four overlapping cohorts receiving 6 days of SB756050 to assess safety, pharmacokinetics, and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 - 60 years of age, inclusive, at the time of signing the informed consent
* A female subject is eligible to participate if she is of non-childbearing potential, defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. FSH and estradiol levels will be checked at Screening for postmenopausal women. Simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<140 pmol/L) is confirmatory.
* Except as noted elsewhere, subjects should have no significant known medical conditions other than T2DM, as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECGs. A subject with a clinical abnormality or laboratory parameters that meets exclusion criteria but is outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* BMI (body mass index) within the range 25-35 kg/m2, inclusive.
* T2DM diagnosed at least 3 months prior to Screening
* Subjects must be treating their T2DM using one of the following regimens: Diet and exercise therapy, Metformin as monotherapy, Sulfonylurea as monotherapy, Metformin and sulfonylurea in combination, DPP-IV inhibitors, either as monotherapy or in combination with other agent(s) on this list at half maximal dose or less, Exenatide, either as monotherapy or in combination with other agent(s) on this list All doses of anti-diabetic medication must have been stable for at least 3 months prior to Screening, and the subject must be willing to wash out from their antidiabetic medications from Day -7 through Day 7.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Has positive pre-study Hepatitis B surface antigen or positive Hepatitis C, result within 3 months of screening. Positive test for HIV antibody. History of uncorrected thyroid dysfunction. ALT and/or AST > 2 times the upper limit of normal at screening. Fasting triglycerides > 450mg/dL at screening. Total Bilirubin > 1.5 times the upper limit of normal at screening. A positive pre-study drug/urine screen and tobacco screen.
* Significant renal disease
* Significant ECG abnormalities
* Systolic pressure > 150 mmHg or <80 mmHg or diastolic blood pressure > 95 mmHg or <60 mmHg at screening.
* Previous use of insulin as a treatment within 3 months of Screening, or for >2 weeks when used for acute illness in the last 12 months prior to Screening, or if used for more than 1 year when associated with GDM.
* Has a history of gastrointestinal disease that could affect absorption within the past year, Gastrointestinal surgery, Chronic or acute pancreatitis.
* History of regular alcohol consumption
* Smoked or used tobacco or nicotine-containing products within the previous 6 months.
* Has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Is taking prohibited medications.
* Unwilling to abstain from caffeine-or xanthine-containing products for 24 hours prior to dosing until Day 7, Use of illicit drugs or nicotine-containing products, Alcohol for 24 hours prior to dosing until Day 7, Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final pharmacokinetic blood samples
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. This includes sensitivity to heparin, if heparin will be used to maintain catheter patency.
* Where participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08-11 (Actual); Primary Completion 2009-03-03 (Actual); Study Completion 2009-03-03 (Actual)

PRIMARY OUTCOMES:
Safety measures including: AEs daily; laboratory testing: day -1,2,5,7 and follow up; ECG: day -1, 2, 5, 6, 7 and follow-up; vital signs: daily; PK parameters day -1,5, and 6. | 6 days of dosing

SECONDARY OUTCOMES:
Pharmacodynamic endpoints will include fasting and meal or OGTT-related weighted mean AUC for glucose, GLP-1 (total and active), glucagon, insulin, PYY (active) and C-peptide levels. | 6 days of dosing
Safety and tolerability parameters including adverse events, clinical laboratory, ECGs and vital signs assessments. | 6 days of dosing
Subject reports of hunger and craving as reported on the Hunger and Craving questionnaire | 6 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Hodge RJ, Lin J, Vasist Johnson LS, Gould EP, Bowers GD, Nunez DJ; SB-756050 Project Team. Safety, Pharmacokinetics, and Pharmacodynamic Effects of a Selective TGR5 Agonist, SB-756050, in Type 2 Diabetes. Clin Pharmacol Drug Dev. 2013 Jul;2(3):213-22. doi: 10.1002/cpdd.34. Epub 2013 May 14. PMID 27121782
- See also: Results for study 111829 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111829?search=study&search_terms=111829#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111829 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register